CLINICAL TRIAL: NCT02977611
Title: The Safety of a High-Dose, Rapid Infusion of Iron Sucrose in a Non-Dialysis Dependent Population
Brief Title: The Safety of a High-Dose, Rapid Infusion of Iron Sucrose
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Clinical Hold
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1611-56
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Dose, Rapid Infusion Iron Sucrose (Experimental): Patients will receive an infusion of 500 mg of iron sucrose over one hour and will be monitored for four hours.
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Iron sucrose — Iron sucrose will be infused at dose of 500 mg over a one hour period
  Other Names: Venofer

SUMMARY:
Iron sucrose infusion is an iron replacement used to treat iron deficiency anemia (not enough iron in the body to make hemoglobin). Iron is a mineral that the body needs to produce hemoglobin, which carries oxygen in the blood. When the body does not get enough iron, it cannot produce enough hemoglobin and you become anemic.

The research study is looking at the side effects of using a higher dose and faster rate of iron sucrose infusion than what is used in standard of care. The purpose of this study is to see if infusion with 500 mg of iron sucrose over a one hour time period can be done safely. If this can be done safely, it may reduce the total number of infusions required and the time for each infusion. This may be less costly and less burdensome to patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient requiring iron infusion

Exclusion Criteria:

* Patients will be excluded from enrollment if they are under the age of 18, unable to give signed consent, are pregnant, have end-stage renal disease, are on hemodialysis (HD), or have a history of clinically significant adverse reactions to iron sucrose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
incidence of adverse events in the study population attributed to drug administration. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Lash, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No